CLINICAL TRIAL: NCT05334212
Title: Evaluating the Impact of Surgical Theater's Patient Engagement 360VR Platform on Spinal Surgery Patient Expectations and Experiences
Brief Title: Impact of Surgical Theater's Patient Engagement
Acronym: ISTPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of support/funding
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20210810
Record Dates: First submitted 2021-11-24; First posted 2022-04-19 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Lumbar Spine Surgeries; Cervical Spine Surgeries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Evaluation of usefulness (Experimental): To evaluate usefulness of Surgical Theater's Patient Engagement 360VR platform in helping align patient expectations and improve patient satisfaction and understanding in spinal surgery consults.
  Interventions: Device: Surgical Theater

INTERVENTIONS:
Device: Surgical Theater — The surgical theater platform uses data from MRI and CT scans, creating a 3d image that can be seen by the patient.

SUMMARY:
To evaluate usefulness of Surgical Theater's Patient Engagement 360VR platform in helping align patient expectations and improve patient satisfaction and understanding in spinal surgery consults.

DETAILED DESCRIPTION:
Surgical Theater is a company that has developed a platform which can be used to describe and explain spinal surgery to patient before they undergo the procedure. The platform specifically implements data from the patient's own MRI and CT scans, creating a 3d reconstruction that can be seen through a virtual reality lens. This technology was developed to help clarify any concerns patient's may have before surgery, and help them better appreciate what will occur in the OR.

Surgical theater has FDA clearance for patient interaction and engagement. Our study is to take surgical theater into our clinics and, after a patient is defined as a surgical candidate, use surgical theater to provide spatial learning and comprehension through modeling so they better understand their surgical plan. Only the SRP system will be used for this study (Surgical Planner).

The intervention is showing surgical theater to patients identified for surgery in clinic routinely. Surgical theater will be offered to all patients offered surgery. No other changes in practice will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-89.
2. Patients undergoing elective lumbar or cervical spine surgeries
3. Those who are receiving Surgical Theater consultation as part of their clinical care

Exclusion Criteria:

1. Age <18 years
2. Non-elective surgery due to emergency, trauma
3. Patients undergoing correction for spinal deformities

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Smith, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University Hospitals at Southwest General Medical Center, Middleburg Heights, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altieri R, Melcarne A, Junemann C, Zeppa P, Zenga F, Garbossa D, Certo F, Barbagallo G. Inferior Fronto-Occipital fascicle anatomy in brain tumor surgeries: From anatomy lab to surgical theater. J Clin Neurosci. 2019 Oct;68:290-294. doi: 10.1016/j.jocn.2019.07.039. Epub 2019 Jul 19. PMID 31331747
- [Background] Bambakidis NC, Selman WR, Sloan AE. Surgical rehearsal platform: potential uses in microsurgery. Neurosurgery. 2013 Oct;73 Suppl 1:122-6. doi: 10.1227/NEU.0000000000000099. PMID 24051875
- [Background] Ehlers JP, Uchida A, Srivastava SK. THE INTEGRATIVE SURGICAL THEATER: Combining Intraoperative Optical Coherence Tomography and 3D Digital Visualization for Vitreoretinal Surgery in the DISCOVER Study. Retina. 2018 Sep;38 Suppl 1(Suppl 1):S88-S96. doi: 10.1097/IAE.0000000000001999. PMID 29256988

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evaluation of Usefulness
Started | 7
Completed | 0
Not Completed | 7
Not completed — Study terminated prematurely | 7

BASELINE CHARACTERISTICS:
Arm/Group | Evaluation of Usefulness
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline EQ-5D Health-Related Quality of Life at 6 Months After Surgery
Description: Reports on 5 dimensions of health: Mobility, Self-care, Usual activities, Pain/Discomfort, Anxiety/Depression. Each score from 1-3 with 1.0 being perfect health.
Time Frame: Visits 1, 2, 3, 4 - 1. Before 360VR consult (Visit 1) 2. Immediately after 360VR consult (Visit 1) 3. Post-op 6 weeks (Visit 2) 4. Post op 3 months (Visit 3) 5. Post op 6 month (Visit 4)
Population: Data not collected
Arm/Group | Evaluation of Usefulness
Number analyzed (Participants) | 0

2. Primary Outcome: Change From Baseline Pain Disability Questionnaire (PDQ) at 6 Months After Surgery
Description: 0-10 Scale to assess how pain affects the ability to function across 15 categories. o 0 (optimal function) to 150 (total disability)
Time Frame: as for outcome 1
Population: Data not collected
Arm/Group | Evaluation of Usefulness
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Patient Satisfaction and Understanding With HCHAPS (Hospital Consumer Assessment of Healthcare Providers and Systems) at 6 Months After Surgery
Description: Understanding - before and after consult, Anxiety level - before and after consult, Satisfaction with consult, HCAHPS - Overall rating of hospital, Satisfied = 9 or 10 rating
Time Frame: as for outcome 1
Population: Data not collected
Arm/Group | Evaluation of Usefulness
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Evaluation of Usefulness
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT05334212/Prot_SAP_001.pdf